CLINICAL TRIAL: NCT00090220
Title: Safety, Immunogenicity, and Efficacy of Gardasil (V501 (Human Papilloma Virus [Types 6, 11, 16, 18] Recombinant Vaccine) in Mid-Adult Women - The FUTURE III (Females United to Unilaterally Reduce Endo/Ectocervical Cancer) Study
Brief Title: A Study to Evaluate the Safety, Immune Response, and Efficacy of Gardasil (V501, qHPV) in Mid-Adult Women (V501-019)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-019; 2004_013
Record Dates: First submitted 2004-08-25; First posted 2004-08-27 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Healthy Adult Female Participants; Prevention; Papillomavirus Infection; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- qHPV Vaccine in Base Study (Experimental): Participants received blinded qHPV vaccination at Day 1, Month 2, and Month 6 of the Base Study
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine
- Placebo in Base Study (Placebo Comparator): Participants received blinded placebo at Day 1, Month 2, and Month 6 in the Base Study. They were eligible to receive open-label qHPV vaccine in Extension 1
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine; Biological: Comparator: Placebo

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine — qHPV intramuscular injection in three 0.5 mL doses over 6 months in the Base Study or EXT1
Biological: Comparator: Placebo — Placebo intramuscular injection in three 0.5 mL doses over 6 months.
  Arms: Placebo in Base Study

SUMMARY:
This study was conducted to assess the safety, immunogenicity, efficacy and long-term effectiveness of a vaccine being evaluated for the prevention of human papillomavirus (HPV) infection and disease in mid-adult women.

DETAILED DESCRIPTION:
The Base study vaccination period (V501-019) encompassed Day 1 through Month 7, during which time participants received randomly assigned, blinded Gardasil™ (V501, qHPV vaccine) or placebo at Day 1, Month 2 and Month 6. The Base study follow-up period continued through approximately Month 48.

The base study was extended in protocol V501-019-10 (EXT1). Participants who received placebo and participants who received only 1 dose of qHPV vaccine in the Base Study were offered a complete, open-label, 3-dose qHPV vaccine regimen (administered at EXT1 Day 1, Month 2 and Month 6). Participants who received only 2 doses of qHPV vaccine in the base study were offered a single additional dose of qHPV vaccine (administered at EXT1 Day 1). Participants were followed to EXT1 Month 7.

A Long Term Follow-Up (LTFU) extension study V501-019-21 (EXT2) was added to observe the long term safety, effectiveness, and immunogenicity of qHPV vaccine in approximately 1,600 women who participated in the Base Study at sites in Colombia. Data were collected over a period of 6-10 years following participant's enrollment in the original Base Study.

ELIGIBILITY:
Inclusion Criteria:

* No history of genital warts, vulvar intraepithelial neoplasia (VIN), or vaginal intraepithelial neoplasia (VaIN)
* Not pregnant and agrees to use effective contraception through Month 7 of the study
* Additional criteria applied

Exclusion Criteria:

* Pregnant
* Concurrently enrolled in a clinical study involving collection of cervical specimens
* Previously received any HPV vaccine
* History of severe allergic reaction that required medical intervention
* Received any immune globulin or blood-derived products within 3 months prior to the first study injection
* History of splenectomy, known immune disorders, or receiving immunosuppressives
* Immunocompromised or diagnosed with human immunodeficiency virus (HIV) infection
* Known thrombocytopenia or any coagulation disorders that could contraindicate intramuscular injections
* History of recent or ongoing alcohol or drug abuse
* Prior treatment for genital warts, VIN, or VaIN
* History of cervical disease (ie, surgical treatment for cervical lesions)
* Hysterectomy

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3819 (Actual)
Dates: Start 2004-06-16 (Actual); Primary Completion 2009-05-21 (Actual); Study Completion 2015-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Munoz N, Manalastas R Jr, Pitisuttithum P, Tresukosol D, Monsonego J, Ault K, Clavel C, Luna J, Myers E, Hood S, Bautista O, Bryan J, Taddeo FJ, Esser MT, Vuocolo S, Haupt RM, Barr E, Saah A. Safety, immunogenicity, and efficacy of quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine in women aged 24-45 years: a randomised, double-blind trial. Lancet. 2009 Jun 6;373(9679):1949-57. doi: 10.1016/S0140-6736(09)60691-7. Epub 2009 Jun 1. PMID 19493565
- [Result] Velicer C, Zhu X, Vuocolo S, Liaw KL, Saah A. Prevalence and incidence of HPV genital infection in women. Sex Transm Dis. 2009 Nov;36(11):696-703. doi: 10.1097/OLQ.0b013e3181ad25ff. PMID 19652630
- [Result] Castellsague X, Munoz N, Pitisuttithum P, Ferris D, Monsonego J, Ault K, Luna J, Myers E, Mallary S, Bautista OM, Bryan J, Vuocolo S, Haupt RM, Saah A. End-of-study safety, immunogenicity, and efficacy of quadrivalent HPV (types 6, 11, 16, 18) recombinant vaccine in adult women 24-45 years of age. Br J Cancer. 2011 Jun 28;105(1):28-37. doi: 10.1038/bjc.2011.185. Epub 2011 May 31. PMID 21629249
- [Result] Luna J, Plata M, Gonzalez M, Correa A, Maldonado I, Nossa C, Radley D, Vuocolo S, Haupt RM, Saah A. Long-term follow-up observation of the safety, immunogenicity, and effectiveness of Gardasil in adult women. PLoS One. 2013 Dec 31;8(12):e83431. doi: 10.1371/journal.pone.0083431. eCollection 2013. PMID 24391768
- [Result] Matys K, Mallary S, Bautista O, Vuocolo S, Manalastas R, Pitisuttithum P, Saah A. Mother-infant transfer of anti-human papillomavirus (HPV) antibodies following vaccination with the quadrivalent HPV (type 6/11/16/18) virus-like particle vaccine. Clin Vaccine Immunol. 2012 Jun;19(6):881-5. doi: 10.1128/CVI.00002-12. Epub 2012 Apr 18. PMID 22518014
- [Result] Garland SM, Ault KA, Gall SA, Paavonen J, Sings HL, Ciprero KL, Saah A, Marino D, Ryan D, Radley D, Zhou H, Haupt RM, Garner EIO; Quadrivalent Human Papillomavirus Vaccine Phase III Investigators. Pregnancy and infant outcomes in the clinical trials of a human papillomavirus type 6/11/16/18 vaccine: a combined analysis of five randomized controlled trials. Obstet Gynecol. 2009 Dec;114(6):1179-1188. doi: 10.1097/AOG.0b013e3181c2ca21. PMID 19935017
- [Derived] Doshi P, Bourgeois F, Hong K, Jones M, Lee H, Shamseer L, Spence O, Jefferson T. Adjuvant-containing control arms in pivotal quadrivalent human papillomavirus vaccine trials: restoration of previously unpublished methodology. BMJ Evid Based Med. 2020 Dec;25(6):213-219. doi: 10.1136/bmjebm-2019-111331. Epub 2020 Mar 17. PMID 32184277
- [Derived] Castellsague X, Ault KA, Bosch FX, Brown D, Cuzick J, Ferris DG, Joura EA, Garland SM, Giuliano AR, Hernandez-Avila M, Huh W, Iversen OE, Kjaer SK, Luna J, Monsonego J, Munoz N, Myers E, Paavonen J, Pitisuttihum P, Steben M, Wheeler CM, Perez G, Saah A, Luxembourg A, Sings HL, Velicer C. Human papillomavirus detection in cervical neoplasia attributed to 12 high-risk human papillomavirus genotypes by region. Papillomavirus Res. 2016 Dec;2:61-69. doi: 10.1016/j.pvr.2016.03.002. Epub 2016 Mar 14. PMID 29074187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Base Study Vaccination Period covers Day 1 to Month 7; Base Study Follow-up Period covers Month 7 up to approximately Month 48; Extension 1 (EXT1) Period covers approximately Month 60 to Month 67; Long-term Follow-up (LTFU, EXT2) covers approximately Month 72 up to Month 120
Groups:
- qHPV Vaccine in Base Study: Participants received Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (qHPV, Gardasil) at Day 1, Month 2, and Month 6
- Placebo in Base Study: Participants received placebo at Day 1, Month 2, and Month 6
- Placebo in Base Study: EXT1: Participants who received placebo in the Base Study were offered open-label qHPV vaccine at EXT1 Day 1 (approximately 60 months after Day 1 of the Base Study), Month 2, and Month 6 and were followed to EXT1 Month 7 (approximately 67 months after Day 1 of the Base Study)
- Incomplete qHPV Regimen in Base Study: EXT1: Participants who received an incomplete regimen of qHPV in the Base Study were offered open-label qHPV vaccine beginning at EXT1 Day 1 (approximately 60 months after Day 1 of the Base Study) and were followed to EXT1 Month 7 (approximately 67 months after Day 1 of the Base Study)
- qHPV Vaccine in Base Study: LTFU (EXT2): Participants at sites in Colombia who received qHPV vaccination in the Base Study were followed from approximately Month 72 up to Month 120 (Year 10) after Day 1 in the Base Study
- Placebo in Base Study and qHPV Vaccine in EXT1: LTFU (EXT2): Participants at sites in Colombia who received placebo or an incomplete regimen of qHPV in the Base Study and open-label qHPV in EXT1 were followed from approximately Month 72 up to Month 120 (Year 10) after Day 1 in the Base Study.
Period: Base Study Vaccination Period
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | Placebo in Base Study: EXT1 | Incomplete qHPV Regimen in Base Study: EXT1 | qHPV Vaccine in Base Study: LTFU (EXT2) | Placebo in Base Study and qHPV Vaccine in EXT1: LTFU (EXT2)
Started | 1911 | 1908 | 0 | 0 | 0 | 0
Vaccinated | 1910 | 1907 | 0 | 0 | 0 | 0
Completed | 1847 | 1845 | 0 | 0 | 0 | 0
Not Completed | 64 | 63 | 0 | 0 | 0 | 0
Not completed — Randomized not Vaccinated | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 24 | 28 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 23 | 27 | 0 | 0 | 0 | 0
Not completed — Patient Moved | 6 | 2 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 4 | 0 | 0 | 0 | 0
Period: Base Study Follow-up Period
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | Placebo in Base Study: EXT1 | Incomplete qHPV Regimen in Base Study: EXT1 | qHPV Vaccine in Base Study: LTFU (EXT2) | Placebo in Base Study and qHPV Vaccine in EXT1: LTFU (EXT2)
Started | 1855 (8 participants did not complete the Vaccination Period but entered the Follow-up Period.) | 1851 (5 participants did not complete the Vaccination Period but entered the Follow-up Period.) | 0 | 0 | 0 | 0
Completed | 1695 | 1687 | 0 | 0 | 0 | 0
Not Completed | 160 | 164 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 88 | 78 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 27 | 36 | 0 | 0 | 0 | 0
Not completed — Patient Moved | 20 | 28 | 0 | 0 | 0 | 0
Not completed — Other | 19 | 21 | 0 | 0 | 0 | 0
Period: Extension 1 (EXT1)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | Placebo in Base Study: EXT1 | Incomplete qHPV Regimen in Base Study: EXT1 | qHPV Vaccine in Base Study: LTFU (EXT2) | Placebo in Base Study and qHPV Vaccine in EXT1: LTFU (EXT2)
Started | 0 | 0 | 1322 (Participation in EXT1 was voluntary; not all participants eligible for EXT1 enrolled.) | 7 (Participation in EXT1 was voluntary; not all participants eligible for EXT1 enrolled.) | 0 | 0
Vaccinated | 0 | 0 | 1321 | 7 | 0 | 0
Completed | 0 | 0 | 1267 | 5 | 0 | 0
Not Completed | 0 | 0 | 55 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 22 | 0 | 0 | 0
Not completed — Moved | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 25 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other reason | 0 | 0 | 2 | 0 | 0 | 0
Period: Long-term Follow-up (EXT2)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | Placebo in Base Study: EXT1 | Incomplete qHPV Regimen in Base Study: EXT1 | qHPV Vaccine in Base Study: LTFU (EXT2) | Placebo in Base Study and qHPV Vaccine in EXT1: LTFU (EXT2)
Started | 0 | 0 | 0 | 0 | 685 (Participation in LTFU was voluntary; not all participants eligible for LTFU enrolled.) | 651 (Participation in LTFU was voluntary; not all participants eligible for LTFU enrolled.)
Completed | 0 | 0 | 0 | 0 | 641 | 623
Not Completed | 0 | 0 | 0 | 0 | 44 | 28
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 38 | 23
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 4
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- qHPV Vaccine in Base Study: Participants received qHPV vaccination at Day 1, Month 2, and Month 6 in the Base Study
- Placebo in Base Study: Participants received placebo at Day 1, Month 2, and Month 6 in the Base Study
- Total: Total of all reporting groups
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | Total
Number analyzed (Participants) | 1911 | 1908 | 3819
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (6.3) | 34.3 (6.3) | 34.3 (6.3)
Age, Continuous [Median (Full Range); unit: Years] — Although the upper age limit for this study was 45 years old, one subject 46 years of age was randomized into the study.
  Years | 35 [24 to 45] | 34 [21 to 46] | 34 [21 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1911 | 1908 | 3819
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 596 | 596 | 1192
  Black | 100 | 82 | 182
  Hispanic American | 822 | 827 | 1649
  Native American | 2 | 1 | 3
  White | 388 | 397 | 785
  Multi-Racial | 3 | 4 | 7
  Polynesian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of HPV 6/11/16/18 Related Persistent Infection, Genital Warts, VIN, VaIN, Vulvar Cancer, Vaginal Cancer, Cervical Dysplasia, Cervical AIS, and Cervical Cancer
Description: The four HPV types were determined by polymerase chain reaction (PCR) testing. VIN = vulvar intraepithelial neoplasia; VaIN = vaginal intraepithelial neoplasia; AIS = adenocarcinoma in situ.
Time Frame: Up to 48 months (4 years) after the first dose of qHPV vaccine in the Base Study
Population: Participants who had no major protocol violations, received all 3 vaccinations, were seronegative to the relevant HPV type at Day 1 and PCR negative to the relevant HPV type Day 1 through Month 7, and provided follow-up data after Month 7
Measure: Number; unit: Incidence per 100 person-years
Groups:
- qHPV in Base Study: Participants received qHPV vaccination at Day 1, Month 2, and Month 6 in the Base Study
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1601 | 1599
Incidence per 100 person-years | 0.2 | 1.7
Statistical Analysis 1: Comparison: qHPV in Base Study vs Placebo in Base Study; Test type: Superiority or Other; Percent Relative Risk Reduction = 88.7, 95% CI [78.1 to 94.8] — Confidence Interval based on binomial tail probabilities and not from a dispersion parameter

2. Primary Outcome: Number of Participants With Vaccine- or Placebo-Related Serious Adverse Events (SAEs) in the Base Study
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse event. A serious adverse event (SAE) is an AE that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs a hospitalization, is a congenital anomaly or birth defect, is a cancer, or is an overdose. Vaccine-related SAEs are those deemed by the investigator to be definitely, probably, or possibly related to study vaccine.
Time Frame: Up to Month 48 (up to 42 months after the third dose of qHPV vaccine in the Base Study)
Population: Participants who received >=1 qHPV vaccination or placebo injection in the Base Study and had safety follow-up
Measure: Number; unit: Participants
Groups:
- Placebo in Base Study: Participants received placebo at Day 1, Month 2, and Month 6 and were followed to Month 48 in the Base Study
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1890 | 1888
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Vaccine-Related SAEs After Vaccine Administration
Description: as for outcome 2
Time Frame: qHPV in Base Study: Up to Month 120; Placebo in Base Study: approximately Month 60 up to Month 120
Population: Participants who received >=1 qHPV vaccination in the Base Study or EXT1 and had safety follow-up
Measure: Number; unit: Participants
Groups:
- Placebo in Base Study: Participants who received placebo or an incomplete qHPV regimen in the Base Study and were offered open-label qHPV vaccine starting at approximately Month 60 in EXT1
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1890 | 1327
Participants | 0 | 1

4. Primary Outcome: Number of Participants With an SAE Resulting in Death After Vaccine Administration
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse event. A serious adverse event (SAE) is an AE that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs a hospitalization, is a congenital anomaly or birth defect, is a cancer, or is an overdose.
Time Frame: qHPV in Base Study: Up to Month 120; Placebo in Base Study: approximately Month 60 up to Month 120
Population: Participants who received >=1 qHPV vaccination in the Base Study or EXT1 and had safety follow-up
Measure: Number; unit: Participants
Groups:
- qHPV in Base Study: All Participants: Participants received qHPV vaccination at Day 1, Month 2, and Month 6 in the Base Study
- Base Study: Placebo: Participants who received placebo or an incomplete qHPV regimen in the Base Study and were offered open-label qHPV vaccine starting at approximately Month 60 in EXT1
Arm/Group | qHPV in Base Study: All Participants | Base Study: Placebo
Number analyzed (Participants) | 1890 | 1327
Participants | 8 | 4

5. Primary Outcome: Cumulative Incidence of HPV 6/11/16/18-related Cervical Intraepithelial Neoplasia (CIN) or Condyloma: Day 1 to Year 4
Description: The four HPV types were determined by PCR testing. Cumulative incidence probability is the probability of becoming an endpoint case at any time from Day 1 to Year 4, conditional on having been event-free at Day 1.
Time Frame: Up to Month 48 (up to 42 months after the third dose of qHPV vaccine in the Base Study)
Population: Participants who had no major protocol violations, received all 3 vaccinations, were seronegative to the HPV types at Day 1 and PCR negative to the HPV types through Month 7, and provided follow-up data.
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Probability
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1602 | 1599
Cumulative Incidence Probability | 0.0006 [0.0001 to 0.0045] | 0.0124 [0.0079 to 0.0195]

6. Primary Outcome: Cumulative Incidence of HPV 6/11/16/18-related CIN or Condyloma: Year 4 to 8
Description: The four HPV types were determined by PCR testing. Cumulative incidence probability is the probability of becoming an endpoint case at any time from Year 4 to Year 8, conditional on having been event-free from Day 1 to Year 4. The analysis windows were cut at the exact time points, e.g., Year 4. Visits and events which occurred after Year 4 due to visit window or follow-up investigations are included in the Year 4 to Year 8 time interval.
Time Frame: From 48 to 96 months (4 to 8 years) after the first dose of qHPV vaccine in the Base Study
Population: Participants who had no major protocol violations, received all 3 vaccinations, were seronegative to the HPV types at Day 1 and PCR negative to the HPV types through Month 7, and provided follow-up data after Year 4. This Outcome Measure applied only to participants who received qHPV in the Base Study.
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Probability
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 927
Cumulative Incidence Probability | 0.0000 [0.0000 to 0.0000]

7. Primary Outcome: Cumulative Incidence of HPV 6/11/16/18-related CIN or Condyloma: Year 6 to 10
Description: The four HPV types were determined by PCR testing. Cumulative incidence probability is the probability of becoming an endpoint case at any time from Year 6 to Year 10, conditional on having been event-free from Day 1 to Year 6.
Time Frame: From 72 to 120 months (6 to 10 years) after the first dose of qHPV vaccine in the Base Study
Population: Participants who had no major protocol violations, received all 3 vaccinations, were seronegative to the HPV types at Day 1 and PCR negative to the HPV types through Month 7, and provided follow-up data after Year 6. This Outcome Measure applied only to participants who received qHPV in the Base Study.
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Probability
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 599
Cumulative Incidence Probability | 0.0000 [0.0000 to 0.0000]

8. Primary Outcome: Incidence Rate of HPV 6/11/16/18-related CIN or Condyloma (Secondary Analysis): Day 1 to Year 4
Description: The four HPV types were determined by PCR testing.
Time Frame: Up to Month 48 (up to 42 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1602 | 1599
Incidence per 100 person-years | 0.0 [0.0 to 0.1] | 0.4 [0.2 to 0.6]

9. Primary Outcome: Incidence Rate of HPV 6/11/16/18-related CIN or Condyloma (Secondary Analysis): Year 4 to 8
Description: The four HPV types were determined by PCR testing. The analysis windows were cut at the exact time points, e.g., Year 4. Visits and events which occurred after Year 4 due to visit window or follow-up investigations are included in the Year 4 to Year 8 time interval.
Time Frame: From 48 to 96 months (4 to 8 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 927
Incidence per 100 person-years | 0.0 [0.0 to 0.2]

10. Primary Outcome: Incidence Rate of HPV 6/11/16/18-related CIN or Condyloma (Secondary Analysis): Year 6 to 10
Description: The four HPV types were determined by PCR testing.
Time Frame: From 72 to 120 months (6 to 10 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 599
Incidence per 100 person-years | 0.0 [0.0 to 0.2]

11. Primary Outcome: Geometric Mean Titer for Anti-HPV Type 6, 11, 16, and 18 Antibody at 1 Month Postdose 3 in the Base Study
Description: Serum antibodies to the HPV Types were determined by Competitive Luminex Immunoassay (cLIA). Geometric Mean Titers (GMT) are reported in milli-Merck Units/mL (mMU/mL). This Outcome Measure evaluated age-specific immunogenicity responses, and applied only to participants who received qHPV in the Base Study.
Time Frame: Month 7 (1 month after the third dose of qHPV vaccine in the Base Study)
Population: Participants who received ≥1 qHPV vaccination. n = participants who were seronegative to the HPV type on Day 1 and PCR negative to the HPV type through Month 7, received 3 doses of qHPV, had a valid postdose 3 serology result for the HPV type, and did not fail any exclusion criteria pertinent to immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- qHPV in Base Study: Participants 24 to 34 Years Old: 24 to 34 year-old participants received qHPV vaccination at Day 1, Month 2, and Month 6 in the Base Study
- qHPV in Base Study: Participants 35 to 45 Years Old: 35 to 45 year-old participants received qHPV vaccination at Day 1, Month 2, and Month 6 in the Base Study
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
mMU/mL
  HPV Type 6: n=1249, 605, 644 | 416.2 [391.9 to 442.0] | 437.4 [401.2 to 476.8] | 397.3 [365.4 to 431.9]
  HPV Type 11: n=1249, 605, 644 | 551.2 [520.5 to 583.6] | 595.1 [548.3 to 646.0] | 512.8 [473.6 to 555.2]
  HPV Type 16: n=1269, 612, 657 | 2225.9 [2101.2 to 2358.0] | 2334.2 [2148.4 to 2536.1] | 2129.5 [1965.7 to 2307.1]
  HPV Type 18: n=1430, 708, 722 | 356.9 [335.8 to 379.4] | 393.1 [360.6 to 428.7] | 324.6 [298.0 to 353.6]

12. Primary Outcome: Geometric Mean Titer for Anti-HPV Type 6, 11, 16, and 18 Antibody at 6 Months Postdose 3 in the Base Study
Description: as for outcome 11
Time Frame: Month 12 (6 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
mMU/mL
  HPV Type 6: n=1225, 589, 636 | 155.1 [147.8 to 162.8] | 157.3 [146.7 to 168.6] | 153.2 [143.3 to 163.8]
  HPV Type 11: n=1225, 589, 636 | 176.9 [168.2 to 186.1] | 184.5 [171.5 to 198.4] | 170.2 [158.6 to 182.5]
  HPV Type 16: n=1236, 588, 648 | 719.6 [684.0 to 757.0] | 743.4 [690.8 to 800.1] | 698.6 [651.3 to 749.2]
  HPV Type 18: n=1387, 678, 709 | 79.2 [74.3 to 84.5] | 84.2 [76.9 to 92.3] | 74.7 [68.3 to 81.7]

13. Primary Outcome: Geometric Mean Titer for Anti-HPV Type 6, 11, 16, and 18 Antibody at 18 Months Postdose 3 in the Base Study
Description: as for outcome 11
Time Frame: Month 24 (18 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
mMU/mL
  HPV Type 6: n=1207, 579, 628 | 70.3 [66.2 to 74.6] | 71.3 [65.4 to 77.8] | 69.3 [63.8 to 75.3]
  HPV Type 11: n=1207, 579, 628 | 77.6 [73.1 to 82.5] | 82.5 [75.6 to 90.0] | 73.4 [67.5 to 79.8]
  HPV Type 16: n=1225, 583, 642 | 278.9 [260.7 to 298.3] | 287.3 [260.6 to 316.9] | 271.4 [247.2 to 297.9]
  HPV Type 18: n=1378, 673, 705 | 28.3 [26.3 to 30.5] | 31.0 [27.9 to 34.4] | 26.0 [23.5 to 28.8]

14. Primary Outcome: Geometric Mean Titer for Anti-HPV Type 6, 11, 16, and 18 Antibody at 30 Months Postdose 3 in the Base Study
Description: as for outcome 11
Time Frame: Month 36 (30 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
mMU/mL
  HPV Type 6: n=1169, 551, 618 | 80.8 [76.4 to 85.5] | 80.5 [74.2 to 87.4] | 81.1 [75.1 to 87.7]
  HPV Type 11: n=1169, 551, 618 | 81.0 [76.6 to 85.6] | 85.3 [78.6 to 92.5] | 77.4 [71.7 to 83.5]
  HPV Type 16: n=1190, 559, 631 | 285.7 [269.0 to 303.4] | 296.2 [271.2 to 323.4] | 276.7 [254.7 to 300.5]
  HPV Type 18: n=1331, 642, 689 | 29.4 [27.4 to 31.6] | 32.2 [29.1 to 35.7] | 27.0 [24.5 to 29.8]

15. Primary Outcome: Geometric Mean Titer for Anti-HPV Type 6, 11, 16, and 18 Antibody at 42 Months Postdose 3 in the Base Study
Description: as for outcome 11
Time Frame: Month 48 (42 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
mMU/mL
  HPV Type 6: n=1152, 536, 616 | 60.9 [57.3 to 64.7] | 59.6 [54.5 to 65.2] | 62.0 [57.1 to 67.4]
  HPV Type 11: n=1152, 536, 616 | 65.9 [62.1 to 69.9] | 69.7 [63.9 to 76.0] | 62.7 [57.8 to 68.0]
  HPV Type 16: n=1172, 544, 628 | 202.1 [189.5 to 215.5] | 213.4 [194.1 to 234.5] | 192.8 [176.5 to 210.5]
  HPV Type 18: n=1313, 625, 688 | 23.1 [21.5 to 24.8] | 25.3 [22.8 to 28.1] | 21.2 [19.2 to 23.4]

16. Primary Outcome: Geometric Mean Titer for Anti-HPV Type 6, 11, 16, and 18 Antibody at 66 Months Postdose 3 in the Base Study
Description: as for outcome 11
Time Frame: Month 72 (66 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- qHPV in Base Study: Participants: Participants received qHPV vaccination at Day 1, Month 2, and Month 6 in the Base Study
- qHPV in Base Study: Participants 24 to 35 Years Old: 24 to 34 year-old participants received qHPV vaccination at Day 1, Month 2, and Month 6 in the Base Study
Arm/Group | qHPV in Base Study: Participants | qHPV in Base Study: Participants 24 to 35 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
mMU/mL
  HPV Type 6: n=468, 198, 270 | 64.3 [58.4 to 70.7] | 60.7 [52.5 to 70.3] | 67.0 [59.1 to 75.9]
  HPV Type 11: n=466, 196, 270 | 64.3 [58.6 to 70.5] | 68.9 [59.7 to 79.5] | 61.1 [54.1 to 69.0]
  HPV Type 16: n=473, 197, 276 | 219.5 [198.3 to 242.9] | 220.3 [188.2 to 257.8] | 218.9 [191.6 to 250.0]
  HPV Type 18: n=530, 237, 293 | 20.9 [18.8 to 23.4] | 22.8 [19.4 to 26.9] | 19.5 [16.8 to 22.6]

17. Primary Outcome: Geometric Mean Titer for Anti-HPV Type 6, 11, 16, and 18 Antibody at 90 Months Postdose 3 in the Base Study
Description: as for outcome 11
Time Frame: Month 96 (90 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | qHPV in Base Study: Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
mMU/mL
  HPV Type 6: n=459, 193, 266 | 56.7 [51.4 to 62.6] | 56.1 [48.2 to 65.3] | 57.2 [50.2 to 65.1]
  HPV Type 11: n=459, 193, 266 | 45.9 [41.7 to 50.6] | 49.6 [42.8 to 57.5] | 43.5 [38.3 to 49.3]
  HPV Type 16: n=464, 192, 272 | 168.3 [151.3 to 187.3] | 174.1 [147.4 to 205.6] | 164.4 [142.9 to 189.0]
  HPV Type 18: n=519, 230, 289 | 18.3 [16.5 to 20.4] | 19.1 [16.3 to 22.4] | 17.7 [15.4 to 20.4]

18. Primary Outcome: Geometric Mean Titer for Anti-HPV Type 6, 11, 16, and 18 Antibody at 114 Months Postdose 3 in the Base Study
Description: as for outcome 11
Time Frame: Month 120 (114 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | qHPV in Base Study: Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
mMU/mL
  HPV Type 6: n=441, 181, 260 | 46.9 [42.2 to 52.0] | 45.7 [38.9 to 53.8] | 47.7 [41.6 to 54.6]
  HPV Type 11: n=441, 181, 260 | 42.3 [38.2 to 46.9] | 45.2 [38.6 to 53.0] | 40.4 [35.4 to 46.2]
  HPV Type 16: n=443, 179, 264 | 140.9 [125.9 to 157.7] | 147.0 [123.2 to 175.5] | 136.9 [118.3 to 158.4]
  HPV Type 18: n=498, 216, 282 | 16.0 [14.3 to 17.8] | 16.6 [14.1 to 19.6] | 15.5 [13.4 to 17.9]

19. Primary Outcome: Percentage of Participants Seropositive for Anti-HPV Antibody at 1 Month Postdose 3 in the Base Study
Description: Serum antibodies to HPV Types 6, 11, 16, and 18 were determined by Competitive Luminex Immunoassay (cLIA). The seropositive thresholds (in mMU/mL) were >20 for Type 6, >16 for Type 11, >20 for Type 16, and >24 for Type 18. This Outcome Measure evaluated age-specific immunogenicity responses, and applied only to participants who received qHPV in the Base Study.
Time Frame: Month 7 (1 month after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
Percentage of participants
  HPV Type 6: n=1249, 605, 644 | 98.4 [97.5 to 99.0] | 98.7 [97.4 to 99.4] | 98.1 [96.8 to 99.0]
  HPV Type 11: n=1249, 605, 644 | 98.1 [97.2 to 98.8] | 98.5 [97.2 to 99.3] | 97.7 [96.2 to 98.7]
  HPV Type 16: n=1269, 612, 657 | 98.8 [98.1 to 99.3] | 99.5 [98.6 to 99.9] | 98.2 [96.8 to 99.1]
  HPV Type 18: n=1430, 708, 722 | 97.3 [96.4 to 98.1] | 98.3 [97.1 to 99.1] | 96.4 [94.8 to 97.6]

20. Primary Outcome: Percentage of Participants Seropositive for Anti-HPV Antibody at 6 Months Postdose 3 in the Base Study
Description: as for outcome 19
Time Frame: Month 12 (6 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
Percentage of participants
  HPV Type 6: n=1225, 589, 636 | 98.7 [97.9 to 99.3] | 98.6 [97.3 to 99.4] | 98.7 [97.5 to 99.5]
  HPV Type 11: n=1225, 589, 636 | 98.8 [98.0 to 99.3] | 99.3 [98.3 to 99.8] | 98.3 [96.9 to 99.1]
  HPV Type 16: n=1236, 588, 648 | 99.7 [99.2 to 99.9] | 99.8 [99.1 to 100] | 99.5 [98.7 to 99.9]
  HPV Type 18: n=1387, 678, 709 | 84.6 [82.6 to 86.5] | 86.1 [83.3 to 88.6] | 83.2 [80.3 to 85.9]

21. Primary Outcome: Percentage of Participants Seropositive for Anti-HPV Antibody at 18 Months Postdose 3 in the Base Study
Description: as for outcome 19
Time Frame: Month 24 (18 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
Percentage of participants
  HPV Type 6: n=1207, 579, 628 | 89.3 [87.4 to 91.0] | 89.5 [86.7 to 91.8] | 89.2 [86.5 to 91.5]
  HPV Type 11: n=1207, 579, 628 | 92.4 [90.7 to 93.8] | 94.0 [91.7 to 95.8] | 90.9 [88.4 to 93.1]
  HPV Type 16: n=1225, 583, 642 | 96.5 [95.3 to 97.4] | 96.9 [95.2 to 98.2] | 96.1 [94.3 to 97.5]
  HPV Type 18: n=1378, 673, 705 | 54.6 [52.0 to 57.3] | 57.4 [53.5 to 61.1] | 52.1 [48.3 to 55.8]

22. Primary Outcome: Percentage of Participants Seropositive for Anti-HPV Antibody at 30 Months Postdose 3 in the Base Study
Description: as for outcome 19
Time Frame: Month 36 (30 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
Percentage of participants
  HPV Type 6: n=1169, 551, 618 | 91.5 [89.8 to 93.1] | 92.0 [89.4 to 94.1] | 91.1 [88.6 to 93.2]
  HPV Type 11: n=1169, 551, 618 | 95.5 [94.1 to 96.6] | 96.7 [94.9 to 98.1] | 94.3 [92.2 to 96.0]
  HPV Type 16: n=1190, 559, 631 | 98.7 [97.9 to 99.3] | 99.1 [97.9 to 99.7] | 98.4 [97.1 to 99.2]
  HPV Type 18: n=1331, 642, 689 | 55.5 [52.8 to 58.2] | 58.7 [54.8 to 62.6] | 52.5 [48.7 to 56.3]

23. Primary Outcome: Percentage of Participants Seropositive for Anti-HPV Antibody at 42 Months Postdose 3 in the Base Study
Description: as for outcome 19
Time Frame: Month 48 (42 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
Percentage of participants
  HPV Type 6: n=1152, 536, 616 | 85.6 [83.4 to 87.6] | 86.2 [83.0 to 89.0] | 85.1 [82.0 to 87.8]
  HPV Type 11: n=1152, 536, 616 | 92.0 [90.3 to 93.5] | 93.8 [91.5 to 95.7] | 90.4 [87.8 to 92.6]
  HPV Type 16: n=1172, 544, 628 | 97.4 [96.3 to 98.2] | 97.8 [96.2 to 98.9] | 97.0 [95.3 to 98.2]
  HPV Type 18: n=1313, 625, 688 | 47.9 [45.2 to 50.6] | 50.7 [46.7 to 54.7] | 45.3 [41.6 to 49.2]

24. Primary Outcome: Percentage of Participants Seropositive for Anti-HPV Antibody at 66 Months Postdose 3 in the Base Study
Description: as for outcome 19
Time Frame: Month 72 (66 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
Percentage of participants
  HPV Type 6: n=468, 198, 270 | 89.1 [85.9 to 91.8] | 89.4 [84.2 to 93.3] | 88.9 [84.5 to 92.4]
  HPV Type 11: n=466, 196, 270 | 92.1 [89.2 to 94.3] | 94.4 [90.2 to 97.2] | 90.4 [86.2 to 93.6]
  HPV Type 16: n=473, 197, 276 | 97.3 [95.3 to 98.5] | 97.5 [94.2 to 99.2] | 97.1 [94.4 to 98.7]
  HPV Type 18: n=530, 237, 293 | 45.3 [41.0 to 49.6] | 48.5 [42.0 to 55.1] | 42.7 [36.9 to 48.5]

25. Primary Outcome: Percentage of Participants Seropositive for Anti-HPV Antibody at 90 Months Postdose 3 in the Base Study
Description: as for outcome 19
Time Frame: Month 96 (96 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
Percentage of participants
  HPV Type 6: n=459, 193, 266 | 84.7 [81.1 to 87.9] | 85.0 [79.1 to 89.7] | 84.6 [79.7 to 88.7]
  HPV Type 11: n=459, 193, 266 | 85.0 [81.4 to 88.1] | 90.7 [85.7 to 94.4] | 80.8 [75.6 to 85.4]
  HPV Type 16: n=464, 192, 272 | 95.5 [93.2 to 97.2] | 95.8 [92.0 to 98.2] | 95.2 [92.0 to 97.4]
  HPV Type 18: n=519, 230, 289 | 40.1 [35.8 to 44.4] | 41.3 [34.9 to 48.0] | 39.1 [33.4 to 45.0]

26. Primary Outcome: Percentage of Participants Seropositive for Anti-HPV Antibody at 114 Months Postdose 3 in the Base Study
Description: as for outcome 19
Time Frame: Month 120 (114 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV in Base Study: All Participants | qHPV in Base Study: Participants 24 to 34 Years Old | qHPV in Base Study: Participants 35 to 45 Years Old
Number analyzed (Participants) | 1910 | 953 | 957
Percentage of participants
  HPV Type 6: n=441, 181, 260 | 78.7 [74.6 to 82.4] | 79.0 [72.3 to 84.7] | 78.5 [73.0 to 83.3]
  HPV Type 11: n=441, 181, 260 | 85.0 [81.4 to 88.2] | 86.7 [80.9 to 91.3] | 83.8 [78.8 to 88.1]
  HPV Type 16: n=443, 179, 264 | 93.9 [91.3 to 95.9] | 95.0 [90.7 to 97.7] | 93.2 [89.4 to 95.9]
  HPV Type 18: n=498, 216, 282 | 35.9 [31.7 to 40.3] | 38.9 [32.3 to 45.7] | 33.7 [28.2 to 39.5]

27. Secondary Outcome: Incidence Rate of HPV 6/11 Related Persistent Infection, Genital Warts, VIN, VaIN, Vulvar Cancer, Vaginal Cancer, Cervical Dysplasia, Cervical AIS, and Cervical Cancer
Description: HPV 6/11: The two types of HPV (types 6/11) were determined by PCR testing
Time Frame: Up to Month 48 (up to 42 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 1
Measure: Number; unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1316 | 1316
Incidence per 100 person-years | 0.0 | 0.9
Statistical Analysis 1: Comparison: qHPV in Base Study vs Placebo in Base Study; Test type: Superiority or Other; Percent Relative Risk Reduction = 94.8, 95% CI [79.9 to 99.4] — Confidence Interval based on binomial tail probabilities and not from a dispersion parameter

28. Secondary Outcome: Cumulative Incidence of HPV 6/11-related Condyloma: Day 1 to Year 4
Description: The four HPV types were determined by PCR testing. Cumulative incidence probability is the probability of becoming an endpoint case at any time from Day 1 to Year 4 conditional on having been event-free at Day 1.
Time Frame: Up to 48 months (4 years) after the first dose of qHPV vaccine or placebo in the Base Study
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Probability
Groups:
- Placebo in the Base Study: Participants received placebo at Day 1, Month 2, and Month 6 in the Base Study
Arm/Group | qHPV in Base Study | Placebo in the Base Study
Number analyzed (Participants) | 1316 | 1316
Cumulative Incidence Probability | 0.0000 [0.0000 to 0.0000] | 0.0055 [0.0026 to 0.0115]

29. Secondary Outcome: Cumulative Incidence of HPV 6/11-related Condyloma: Year 4 to Year 8
Description: The four HPV types were determined by PCR testing. Cumulative incidence probability is the probability of becoming an endpoint case at any time from Year 4 to Year 8 conditional on having been event-free from Day 1 to Year 4. The analysis windows were cut at the exact time points, e.g., Year 4. Visits and events which occurred after Year 4 due to visit window or follow-up investigations are included in the Year 4 to Year 8 time interval.
Time Frame: From 48 to 96 months (4 to 8 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Probability
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 751
Cumulative Incidence Probability | 0.0000 [0.0000 to 0.0000]

30. Secondary Outcome: Cumulative Incidence of HPV 6/11-related Condyloma: Year 6 to Year 10
Description: The four HPV types were determined by PCR testing. Cumulative incidence probability is the probability of becoming an endpoint case at any time from Year 6 to Year 10 conditional on having been event-free from Day 1 to Year 6.
Time Frame: From 72 to 120 months (6 to 10 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Probability
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 492
Cumulative Incidence Probability | 0.0000 [0.0000 to 0.0000]

31. Secondary Outcome: Incidence Rate of HPV 6/11-related Condyloma (Secondary Analysis): Day 1 to Year 4
Description: The four HPV types were determined by PCR testing.
Time Frame: Up to 48 months (4 years) after the first dose of qHPV vaccine or placebo in the Base Study
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study | Placebo in the Base Study
Number analyzed (Participants) | 1316 | 1316
Incidence per 100 person-years | 0.0 [0.0 to 0.1] | 0.2 [0.1 to 0.3]

32. Secondary Outcome: Incidence Rate of HPV 6/11-related Condyloma (Secondary Analysis): Year 4 to Year 8
Description: as for outcome 9
Time Frame: From 48 to 96 months (4 to 8 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 751
Incidence per 100 person-years | 0.0 [0.0 to 0.2]

33. Secondary Outcome: Incidence Rate of HPV 6/11-related Condyloma (Secondary Analysis): Year 6 to Year 10
Description: as for outcome 30
Time Frame: From 72 to 120 months (6 to 10 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 492
Incidence per 100 person-years | 0.0 [0.0 to 0.2]

34. Secondary Outcome: Incidence Rate of HPV 31/33/35/52/58 Related Persistent Infection, Genital Warts, VIN, VaIN, Vulvar Cancer, Vaginal Cancer, Cervical Dysplasia, Cervical AIS, and Cervical Cancer
Description: This outcome measure was not analyzed because of diminished interest by experts in composite efficacy endpoints associated with these HPV types
Time Frame: Up to Month 48 (up to 42 months after the third dose of qHPV vaccine in the Base Study)
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 0 | 0

35. Other Pre Specified Outcome: Incidence Rate of HPV 16/18 Related Persistent Infection, Genital Warts, VIN, VaIN, Vulvar Cancer, Vaginal Cancer, Cervical Dysplasia, Cervical AIS, and Cervical Cancer
Description: HPV 16/18: The two types of HPV (types 16/18) were determined by PCR testing
Time Frame: Up to Month 48 (up to 42 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 1
Measure: Number; unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1587 | 1571
Incidence per 100 person-years | 0.2 | 1.0
Statistical Analysis 1: Comparison: qHPV in Base Study vs Placebo in Base Study; Test type: Superiority or Other; Percent Relative Risk Reduction = 84.7, 95% CI [67.5 to 93.7] — Confidence Interval based on binomial tail probabilities and not from a dispersion parameter

36. Other Pre Specified Outcome: Cumulative Incidence of HPV 16/18-related CIN 2 or Worse: Day 1 to Year 4
Description: as for outcome 28
Time Frame: Up to Month 48 (up to 42 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Probability
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1570 | 1558
Cumulative Incidence Probability | 0.0007 [0.0001 to 0.0046] | 0.0041 [0.0019 to 0.0092]

37. Other Pre Specified Outcome: Cumulative Incidence of HPV 16/18-related CIN 2 or Worse: Year 4 to 8
Description: as for outcome 29
Time Frame: From 48 to 96 months (4 to 8 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Probability
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 842
Cumulative Incidence Probability | 0.0000 [0.0000 to 0.0000]

38. Other Pre Specified Outcome: Cumulative Incidence of HPV 16/18-related CIN 2 or Worse: Year 6 to 10
Description: as for outcome 30
Time Frame: From 72 to 120 months (6 to 10 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Probability
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 541
Cumulative Incidence Probability | 0.0000 [0.0000 to 0.0000]

39. Other Pre Specified Outcome: Incidence Rate of HPV 16/18-related CIN 2 or Worse (Secondary Analysis): Day 1 to Year 4
Description: The four HPV types were determined by PCR testing.
Time Frame: Up to Month 48 (up to 42 months after the third dose of qHPV vaccine in the Base Study)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1570 | 1558
Incidence per 100 person-years | 0.0 [0.0 to 0.1] | 0.1 [0.0 to 0.3]

40. Other Pre Specified Outcome: Incidence Rate of HPV 16/18-related CIN 2 or Worse (Secondary Analysis): Year 4 to 8
Description: as for outcome 9
Time Frame: From 48 to 96 months (4 to 8 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 842
Incidence per 100 person-years | 0.0 [0.0 to 0.2]

41. Other Pre Specified Outcome: Incidence Rate of HPV 16/18-related CIN 2 or Worse (Secondary Analysis): Year 6 to 10
Description: The four HPV types were determined by PCR testing.
Time Frame: From 72 to 120 months (6 to 10 years) after the first dose of qHPV vaccine in the Base Study
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | qHPV in Base Study
Number analyzed (Participants) | 541
Incidence per 100 person-years | 0.0 [0.0 to 0.2]

ADVERSE EVENTS:
Time Frame: Base study: all AEs Day 1 to approximately Month 48; EXT1: SAEs only approximately Month 60 to Month 67; LTFU (EXT2): SAEs only approximately Month 72 to Month 120. Other AEs were not solicited in EXT1 or LTFU (EXT2).
Description: Base Study: MedDRA v12.0; EXT1: MedDRA v14.1; LTFU (EXT2): MedDRA v18.1.
  Adverse events are reported for all participants who received ≥1 dose of qHPV or placebo and had safety follow-up data.
  Although other AEs were not solicited in EXT1 and LTFU (EXT2), some were voluntarily reported.
Groups:
- qHPV Vaccine: Base Study: Participants received qHPV vaccination at Day 1, Month 2, and Month 6 and were followed up to approximately Month 48
- Placebo: Base Study: Participants received placebo at Day 1, Month 2, and Month 6 and were followed up to approximately Month 48
- qHPV Vaccine: EXT1: Participants who received placebo or an incomplete regimen of qHPV in the Base Study were offered open-label qHPV vaccine starting at approximately Month 60 (EXT1) and were followed up to Month 67
- Long-term Follow-up: EXT2: Participants at sites in Colombia who received qHPV vaccination in the Base Study or in EXT1 were followed from Month 72 up to approximately Month 120 in LTFU (EXT2)
Arm/Group | qHPV Vaccine: Base Study | Placebo: Base Study | qHPV Vaccine: EXT1 | Long-term Follow-up: EXT2
Serious Adverse Events (participants affected / at risk) | 15/1890 | 17/1888 | 6/1327 | 6/1336
Other Adverse Events (participants affected / at risk) | 1565/1890 | 1390/1888 | 2/1327 | 0/1336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV Vaccine: Base Study (N=1890) | Placebo: Base Study (N=1888) | qHPV Vaccine: EXT1 (N=1327) | Long-term Follow-up: EXT2 (N=1336)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Peritoneal tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis gastrointestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gestational trophoblastic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
False labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fallopian tube cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV Vaccine: Base Study (N=1890) | Placebo: Base Study (N=1888) | qHPV Vaccine: EXT1 (N=1327) | Long-term Follow-up: EXT2 (N=1336)
Injection site erythema (General disorders) | 275 (392) | 200 (280) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1424 (3168) | 1173 (2252) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 356 (530) | 215 (293) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 219 (295) | 232 (298) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 98 (107) | 101 (113) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 528 (857) | 519 (787) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication or presentation